CLINICAL TRIAL: NCT05086809
Title: BC109 - Investigation of an Updated Bone-anchored Sound Processor
Brief Title: Investigation of an Updated Bone-anchored Sound Processor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: BC109
Record Dates: First submitted 2021-09-27; First posted 2021-10-21 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2021-10

CONDITIONS: Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Mixed; Hearing Disorders; Deafness; Ear Diseases; Otorhinolaryngologic Diseases; Sensation Disorders; Neurologic Manifestations; Nervous System Diseases
Keywords: BAHS; Ponto
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Hearing Disorders; Deafness; Ear Diseases; Otorhinolaryngologic Diseases; Sensation Disorders; Neurologic Manifestations; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: The study includes four laboratory visits and three field trial periods. The first trial period is included to ensure a homogenous baseline. After the first trial period, the study is designed as a two-period, two-sequence crossover trial to compare two sound processors (Device A & Device B). Each participant is randomized into one of two sequences: (1) Device A then B, or (2) Device B then A, such that (about) half of the participants are assigned to one sequence and the other half to the second sequence.
Who Masked: Participant
Masking Description: The participants are blinded to the tested conditions in the lab, used for assessment of the primary objective, but the participants are not blinded to the sound processors used during the three trial periods, due to different appearance of the sound processors, making it possible to distinguish between the sound processors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AAB (Active Comparator): Starts with Device A in first and second trial period and change to Device B in third trial period.
  Interventions: Device: Device A; Device: Device B
- ABA (Active Comparator): Starts with Device A in first trial period, wears Device B in second trial period and change to Device A in third trial period.
  Interventions: Device: Device A; Device: Device B

INTERVENTIONS:
Device: Device A — Participant wear Device A and evaluate the performance of the device.
Device: Device B — Participant wear Device B and evaluate the performance of the device.

SUMMARY:
The study is a prospective, single-center, comparative, cross-over study with within-subject control design. In the investigation an updated sound processor will be tested at compared to the CE marked Ponto 3 SuperPower sound processor (available on the market since December 2016) in order to establish marketing claim(s) on the updated sound processor.

The performance of the two sound processors will be evaluated via speech and hearing tests, and patient reported outcomes.

DETAILED DESCRIPTION:
The investigation is a premarket investigation with the purpose of gathering knowledge on the performance of an updated sound processor compared to the CE marked Ponto 3 SuperPower sound processor to establish marketing claim(s) on the updated sound processor.

The recruitment for this clinical investigation will be performed among subjects who have already received a Ponto 3 SuperPower sound processor as a minimum three month prior to the study. 12-15 adult Ponto 3 SuperPower users with a conductive, mixed hearing loss or single-sided deafness will be included.

The study is a prospective, single-center, comparative, cross-over study with within-subject control design. The study includes four laboratory visits and three field trial periods. After the first trial period, which is included to ensure a homogenous baseline, the study is designed as a two-period, two-sequence crossover trial to compare the two sound processors (Device A & Device B). Each participant is randomized into one of two sequences: (1) Device A then B, or (2) Device B then A, such that (about) half of the participants are assigned to one sequence and the other half to the second sequence.

This study is designed to combine audiological assessments (hearing and speech tests) in the laboratory and subjective self-reported outcomes collected during and after field trial periods with the investigational device and the comparator device (Ponto 3 SuperPower). The primary outcome of this study is to demonstrate that Open Sound Navigator in the updated sound processor provides subjects with improved speech recognition in noise.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Adult subjects (18 years or older)
3. Subjects using a Ponto 3 SuperPower on Oticon Medical compatible abutment
4. Experienced BAHS users with a minimum experience of 3 months.
5. Subjects with:

   1. conductive or mixed hearing loss with pure tone average (PTA) bone conduction (BC) threshold (measured at 0.5, 1, 2 and 3 kHz) of the indicated ear better than or equal to 65 dB HL as measured in situ with Ponto 3 SuperPower at Visit 1.
   2. OR subjects who have a profound sensorineural hearing loss in one ear and normal hearing in the opposite ear (i.e., SSD). The pure tone average (PTA) air conduction (AC) threshold of the hearing ear should then be better than or equal to 20 dB HL (measured at 0.5, 1, 2 and 3 kHz) as reported in the patient's Noah file.
   3. OR subjects who are indicated for an air-conduction contralateral routing of signals (AC CROS) hearing aid, but who for some reason cannot or will not use an AC CROS (as per investigator discretion).
6. Fluent in Danish

Exclusion Criteria:

Subjects meeting any of the following criteria will not be permitted to participate in the investigation:

1. Known abnormally progressive BC hearing loss as judged by the investigator
2. Subjects with known mixed losses where the sensorineural part of the hearing loss is of retro-cochlear or central origin
3. Participation in another clinical investigation which might cause interference with study participation.
4. Subjects who do not have the ability or are un-willing to follow investigational procedures/requirements, e.g. to complete questionnaires, according to investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
To demonstrate that OSN in Device A provides subjects with improved speech recognition in noise. | 4 weeks or 6 weeks
  Difference in signal-to-noise ratio at 70% correct (referred to as SRT70) between OSN OFF and OSN ON after field trial with Device A (incl. automatics).

SECONDARY OUTCOMES:
To assess the preference of BAHS sound processor. | 6 weeks
  Percentage (%) of subjects who prefer Device A over Device B in noisy sound environments.
To assess the improvement of hearing with Device A. | Baseline
  1. Functional gain with Device A, i.e. the difference in dB between unaided and aided sound field thresholds, for frequencies 250, 500, 1000, 2000, 3000, 4000, 6000 and 8000 Hz.
  2. Functional gain with Device A, see definition above, calculated on average for frequencies 500, 1000, 2000 and 4000 Hz (PTA4).
To assess the degree to which Device A compensates for the BC hearing loss for the group CHL/MHL | Baseline
  1. Effective gain defined as the difference in dB between aided sound field thresholds with Device A, and BC in-situ thresholds on the aided ear(s). The effective gain is calculated for frequencies 250, 500, 1000, 2000, 3000, 4000, 6000 and 8000 Hz.
  2. Effective gain with Device A, see definition above, calculated in average for frequencies 500, 1000, 2000 and 4000 Hz (PTA4).
To assess the improvement in speech recognition with Device A in quiet. | 2 weeks
  Difference in speech recognition score in percent between unaided and aided, assessed in quiet on the aided ear(s).
To assess performance in speech recognition in noise with Device A and Device B in Omni settings. | Baseline
  Difference in SRT70 between Device A and Device B in Omni settings as measured at Visit 1.
To assess the improvement in speech recognition in noise with Device B in full directional settings as compared to omnidirectional. | 4 weeks or 6 weeks
  Difference in signal-to-noise ratio at 70% correct (referred to as SRT70) between Omni and Full Dir after field trial with Device B.
To compare the improvement in speech recognition in noise with OSN ON in Device A (re Omni) with the improvement of full directionality in Device B (re Omni). | 4 weeks or 6 weeks
  Comparison of the difference in SRT70 between OSN OFF vs. OSN ON in Device A and Omni vs. Full Dir in Device B.
To assess self-reported performance with Device A and Device B. | 4 weeks or 6 weeks
  1. Average SSQ12 scores with Device A for each question, sub-scales and in total.
  2. Average SSQ12 scores with Device B for each question, sub-scales and in total.
  3. Difference in SSQ12 scores between Device A and Device B for each question, sub-scales and in total.
To assess self-reported ratings of sound quality, speech intelligibility, and overall performance with Device A and Device B. | 1 week, 4 weeks and 6 weeks
  1. Average ratings with Device A for each question of the "SPSK sound quality" questionnaire completed during the 1. field trial with Device A as obtained via phone interview
  2. Average ratings with Device A for each question of the "SPSK sound quality" questionnaire completed during the 2. or 3. field trial with Device A
  3. Average ratings with Device B for each question of the "SPSK sound quality" questionnaire completed during the 2. or 3. field trial with Device B
  4. Difference in ratings between Device A and Device B for each question of the "SPSK sound quality" questionnaire
  5. Average ratings with Device A for each question of the "SPSK situations" questionnaire completed during the 2. or 3. field trial with Device A
  6. Average ratings with Device B for each question of the "SPSK situations" questionnaire completed during the 2. or 3. field trial with Device B
  7. Difference in ratings between Device A and Device B for each question of the "SPSK situations" questionnaire
To assess the difference in BC thresholds as measured in-situ with Device A and via conventional BC audiometry. | Baseline and 2 weeks
  Difference in dB between BC in situ thresholds and BC thresholds measured with conventional BC audiometry.
To assess the difference in BC thresholds as measured in-situ with Device A and Device B. | Baseline
  Difference in dB between BC in situ thresholds measured with Device A and Device B.
To confirm the safety profile of the Device A in terms of the occurrence of adverse events and serious adverse events. | 1 week, 2 weeks, 4 weeks and 6 weeks
  Tabulated adverse events and serious adverse event related to the Device A reported throughout the study.

OTHER OUTCOMES:
To assess the improvement in speech recognition in noise with Device A with OSN ON vs. OSN OFF as a function of hearing loss. | Baseline and week 4 or week 6
  Correlation of the difference between OSN OFF and OSN ON after field trial with Device A (incl. automatics) and PTA4 BC in situ for subjects with SSD and subjects with conductive/mixed hearing loss.
To list comments and reactions from the subjects with Device A and Device B. | Baseline, 2 weeks and 4 weeks
  Immediate reactions collected with each sound processor before field trial.
To list comments and reactions from the subjects with Device A and Device B. | 2 weeks
  Comments on any difference between phone interview and subject's feedback collected at V2 after first field trial with Device A (without automatics).
To assess usage of device for each field trial period. | 2 weeks, 4 weeks and 6 weeks
  Average hours of usage of each sound processor for each field trial.
To assess usage of device and batteries for each field trial period. | 2 weeks, 4 weeks and 6 weeks
  Frequency of battery replacement for each sound processor for each field trial.

CONTACTS AND LOCATIONS:
Overall Officials: Mona El Hichou, MSc, Principal Investigator — Oticon Medical c/o Oticon A/S
Locations (1):
- Oticon Medical c/o Oticon A/S, Copenhagen, Smørum, Denmark